CLINICAL TRIAL: NCT00501722
Title: SR121463B in Cirrhotic Ascites Treatment With Hyponatraemia: A Placebo-Controlled, Dose-Comparison Study
Brief Title: Satavaptan Dose-Ranging Study in Hyponatraemic Patients With Cirrhotic Ascites
Acronym: Hypo~CAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI4521; LTS5634; LTS10209
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Ascites; Liver Cirrhosis
Keywords: cirrhotic ascites; hyponatraemia
MeSH Terms: conditions — Ascites; Liver Cirrhosis; Hyponatremia | interventions — satavaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: satavaptan (SR121463B)

SUMMARY:
The primary objective is to determine the optimal dose or range of doses of SR121463B for the treatment of ascites and the correction of hyponatraemia when used concomitantly with a standard dose regimen of spironolactone.

The secondary objective is to determine the tolerability of different fixed doses of SR121463B over a 14 day treatment period in cirrhotic ascites.

This Hypo~CAT study is followed by a single-blind, placebo-controlled, one-year long-term safety extension (Expo~CAT). The first extension is followed by another long-term study (PASCCAL-1).

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of the liver confirmed by ultrasound, endoscopic examination, or biochemical evidence
* Moderate or tense ascites
* Patients with hyponatremia, defined as a serum sodium concentration of ≤130 mmol/L

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-04; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
change in body weight, change in serum sodium | within 14 days

SECONDARY OUTCOMES:
abdominal girth and discomfort | 14 days
paracentesis | 14 days
trail-making test and quality of life | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (13):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Barcelona, Spain

REFERENCES:
- [Derived] Gines P, Wong F, Watson H, Milutinovic S, del Arbol LR, Olteanu D; HypoCAT Study Investigators. Effects of satavaptan, a selective vasopressin V(2) receptor antagonist, on ascites and serum sodium in cirrhosis with hyponatremia: a randomized trial. Hepatology. 2008 Jul;48(1):204-13. doi: 10.1002/hep.22293. PMID 18508290
- See also: Related Info — http://www.sanofi-aventis.com